CLINICAL TRIAL: NCT03700034
Title: A Cluster-randomized Trial of an mHealth Integrated Model of Hypertension, Diabetes and Antenatal Care in Primary Care Settings in India and Nepal
Brief Title: mHealth Integrated Model of Hypertension, Diabetes and Antenatal Care in India and Nepal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Public Health Foundation of India (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dorairaj Prabhakaran, Vice President - Research and Policy, Public Health Foundation of India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CTRI/2019/01/016857
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Gestational Diabetes Mellitus (GDM); Pregnancy Induced Hypertension (PIH); Anemia
Keywords: Antenatal care; Pregnancy care; Pregnancy complications; Pregnancy Induced Hypertension; Gestational Diabetes Mellitus; Anemia
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced; Anemia; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth integrated model of hypertension, diabetes, anemia, and antenatal care (Experimental): The mIRA trial intervention will consist of an electronic decision support system (EDSS), provided to healthcare providers at primary-level facilities in India and Nepal to deliver enhanced ANC with improved detection and management of pregnancy-induced hypertension (PIH), gestational diabetes mellitus (GDM) and anemia.
  Interventions: Other: mHealth Integrated Model of Antenatal Care
- Routine antenatal care (No Intervention): In the control clusters, pregnant women will receive the existing standard of care (usual care) from Frontline Health Workers (FHWs). Evidence-based guidelines in the form of posters/pamphlets on current national and state guidelines on screening and management of pregnancy-induced hypertension (PIH), gestational diabetes mellitus (GDM), anemia, and routine ANC procedures will be provided to all the control health facilities.

INTERVENTIONS:
Other: mHealth Integrated Model of Antenatal Care — In the intervention facilities, antenatal care (ANC) will be provided to all pregnant women using the mIRA electronic decision support system (EDSS) by ANMs (Auxiliary Nurse Midwife), Staff nurses, or Medical Officers (MOs). These frontline healthcare workers (FHWs) will be trained to use the EDSS and will also be provided "refresher" training on the guideline-recommended processes of ANC. This training will enable them to use the mIRA EDSS in the provision of ANC. Non-physician FHWs (ANMs and staff nurses) will screen, detect, and refer PIH, GDM, and severe anemia cases. They will not prescribe treatments, but will carry out all other duties including diagnosis, referral to the MO to prescribe drugs, provide lifestyle advice, follow-up, and subsequently support adherence to management plans.
  Other Names: Electronic Decision Based System (EDSS)
  Arms: mHealth integrated model of hypertension, diabetes, anemia, and antenatal care

SUMMARY:
Our research aims to address a critical gap in the provision of quality antenatal care (ANC) in India and Nepal, by developing and evaluating an intervention comprising of a tablet-based electronic decision support system (EDSS). This intervention -"mIRA" - is an mHealth integrated model of hypertension, diabetes, and antenatal care in primary care settings. mIRA aims to (a) prompt frontline health workers (FHWs) to provide evidence-based routine ANC, and also enhance the detection and management of Pregnancy Induced Hypertension (PIH), Gestational Diabetes Mellitus (GDM), and anemia, whilst improving adherence to National ANC guidelines; (b) facilitate record-keeping and reporting and; (c) link providers across various levels of care to improve continuity of care.

A cluster randomized controlled (cRCT) to assess the effectiveness of the mIRA EDSS in improving ANC and enhancing the detection and management of Pregnancy Induced Hypertension (PIH), Gestational Diabetes Mellitus (GDM), and anemia will be conducted in Telangana, India. A mixed-methods process evaluation will be conducted in both India and Nepal. The process evaluation will contribute to our understanding of the mechanisms contributing to changes (improvement) in the quality of ANC by using the EDSS intervention.

DETAILED DESCRIPTION:
The cRCT aims to evaluate the effectiveness of a tablet-based EDSS in improving the quality of ANC and enhancing the detection and management of PIH, GDM, and anemia at primary care level health facilities in five districts of Telangana State: Medak, Rangareddy, Siddipet, Vikarabad, and Yadadri Bhuvangiri. The EDSS will use evidence-based algorithms to suggest recommendations to the FHWs for providing ANC, based on the pregnant woman's history, examination, and investigations, as well as incorporate reminders to ensure all relevant components of ANC are recorded. The aim is to ensure that ANC components received during multiple visits from multiple healthcare providers are captured and contribute to coordinated care. FHWs, primarily Auxiliary Nurse Midwives (ANMs), will use the EDSS during ANC consultations with pregnant women at Sub-Centres, while at the Primary Health Centres (PHCs), this will be used by Medical Officers (MOs) and staff nurses.

In these selected districts, which are predominantly rural, 66 clusters with each cluster comprising a PHC and its two reporting Sub-Centres, will be randomized with a 1:1 allocation ratio to the intervention arm (providing ANC using the mIRA EDSS intervention) and the control arm (providing usual care), using a computer-generated randomization schedule stratified by the district. Covariate constrained randomization will be used to balance the arms on the following baseline covariates: the presence of a laboratory and laboratory technician (yes/no); more than three staff providing ANC (yes/no); facility type (PHCs that are open 24/7 or those not open 24/7).

The cRCT will not be conducted In Nepal, however, the mIRA EDSS will be implemented at government Health Posts (HP), government Primary Health Care Centers (PHCCs), and Dhulikhel Hospital Outreach Centers (DHORCs), in four catchment districts (Kavrepalanchok, Sindhupalchowk, Sindhuli, and Dolakha) of Dhulikhel Hospital. A pre-post EDSS implementation outcome evaluation will be conducted. The process evaluation research activities conducted in India and Nepal will be the same (including a baseline facility survey, routine monitoring, and audit of record-keeping), except for a longitudinal case study and a time-motion study that will be conducted only in Nepal. Additionally, endline qualitative in-depth interviews with healthcare providers, facility managers, district and state health officials and policymakers, and with members of the Public Health Foundation of India team (intervention implementors) will be conducted only in India.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women visiting a trial facility up to the end of the 28th week of gestation
* Women who are planning to remain within the five study districts until at least one-month post-partum OR women whose mothers reside in the selected districts

Exclusion Criteria:

• Women coming to the trial facility for a non-routine ANC visit (for example, to get a laboratory investigation, to collect a report or her medicine)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1320 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Mean number of four selected ANC components delivered by the healthcare providers per visit, observed over two visits- the trial enrolment visit and the next routine ANC appointment. | Up to 28 weeks of gestation till the study completion with an average follow-up period of 3 months
  This will be a composite score calculated as per the performance of the number of selected ANC components delivered or completed by the healthcare provider. The four selected components are: 1) the measurement and recording of systolic and diastolic blood pressure; 2) measurement of blood glucose, 3) performing urinary dipstick test for proteinuria and 4) conducting hemoglobin tests. The action of completing each of the aforementioned components by the healthcare provider will count as a score of one. Thus, completion of all four components will account to a score of four.

SECONDARY OUTCOMES:
Mean number of the four selected ANC components delivered by the healthcare provider observed at the trial enrolment visit | Up to 28 weeks of gestation
  This will be a composite score calculated as per the performance of the number of selected ANC components delivered or completed by the healthcare provider. The four selected components are: 1) the measurement and recording of systolic and diastolic blood pressure; 2) measurement of blood glucose, 3) performing urinary dipstick test for proteinuria and 4) conducting hemoglobin tests. The action of completing each of the aforementioned components by the healthcare provider will count as a score of one. Thus, completion of all four components will account to a score of four.
Mean number of the current pregnancy symptoms discussed with participants (either by the provider asking or the woman mentioning), observed over the two visits. | Up to 28 weeks of gestation till the study completion with an average follow-up period of 3 months
  Symptoms include: nausea, vomiting, vaginal bleeding, severe headache, decreased or absent fetal movement, severe abdominal pain, blurred vision
Proportion of providers who took the appropriate action (as defined by the EDSS) in response to aforementioned current pregnancy symptoms or who were told that they had hypertension in pregnancy, GDM or anemia | Up to 28 weeks of gestation till the study completion with an average follow-up period of 3 months
  Symptoms for which a response is expected from the provider: vomiting, vaginal bleeding, severe headache, decreased or absent foetal movement, severe abdominal pain or blurred vision or who were told that they had hypertension in pregnancy, GDM or anemia
Mean number of the danger signs mentioned to each participant by the healthcare provider for which she is advised to return for help | Up to 28 weeks of gestation till the study completion with an average follow-up period of 3 months
  Danger signs include severe vomiting, vaginal bleeding, severe headache, decreased or no foetal movement, severe abdominal pain, blurred vision
Proportion of participants with clinical parameters indicative of PIH, GDM or severe anemia | Up to 28 weeks of gestation till the study completion with an average follow-up period of 3 months
  Conditions diagnosed as: hypertension (SBP≥ 140 mmHg and DBP≥90 mmHg), GDM (venous blood glucose: fasting >92 mg/dL, 1 h OGTT (Oral Glucose Tolerance Test) >180 mg/dL, 2 h OGTT >153-199 mg/dL; glucometer test values: fasting >92 mg/dL, 1 h OGTT >198 mg/dL, 2 h OGTT >168 mg/dL) or severe anemia (<7g/dL)
Proportion of participants who were told by the provider that they had PIH, GDM or severe anemia | Up to 28 weeks of gestation till the study completion with an average follow-up period of 3 months
  Conditions diagnosed as: hypertension (SBP≥ 140 mmHg and DBP≥90 mmHg), GDM (venous blood glucose: fasting >92 mg/dL, 1 h OGTT (Oral Glucose Tolerance Test) >180 mg/dL, 2 h OGTT >153-199 mg/dL; glucometer test values: fasting >92 mg/dL, 1 h OGTT >198 mg/dL, 2 h OGTT >168 mg/dL) or severe anemia (<7g/dL)
Mean number of quality antenatal care components delivered in the enrolment visit | Up to 28 weeks of gestation
  The components are as follows:
  tests completed: blood pressure; blood glucose; urinary dipstick; hemoglobin tests
  Provider:
  symptom check: nausea; vomiting; vaginal bleeding; severe headache, decreased or absent foetal movement, severe abdominal pain, blurred vision
  warning about: severe vomiting; vaginal bleeding; severe headache; decreased or no foetal movement: severe abdominal pain; blurred vision
  counseling on diet
  enquiring about mental health
  recording ANC related information on the women-held MCP (Maternal and Chlid Protection) card

CONTACTS AND LOCATIONS:
Overall Officials: Dorairaj Prabhakaran, DM, Principal Investigator — Vice President, Research and Policy
Locations (6):
- India (5):
  - Primary Health Centres (PHCs), Medak, Telangana
  - Primary Health Centres (PHCs), Rangareddy, Telangana
  - Primary Health Centres, Siddipet, Telangana
  - Primary Health Centres (PHCs), Vikārābād, Telangana
  - Primary Health Centres (PHCs), Yadadri Bhuvnagiri, Telangana
- Health posts, Dhulikhel, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohan S, Chaudhry M, McCarthy O, Jarhyan P, Calvert C, Jindal D, Shakya R, Radovich E, Kondal D, Penn-Kekana L, Basany K, Roy A, Tandon N, Shrestha A, Shrestha A, Karmacharya B, Cairns J, Perel P, Campbell OMR, Prabhakaran D. A cluster randomized controlled trial of an electronic decision-support system to enhance antenatal care services in pregnancy at primary healthcare level in Telangana, India: trial protocol. BMC Pregnancy Childbirth. 2023 Jan 26;23(1):72. doi: 10.1186/s12884-022-05249-y. PMID 36703109